CLINICAL TRIAL: NCT01705574
Title: A Randomized, Double-blind Phase 3B Study to Evaluate the Safety and Efficacy of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate Versus Ritonavir-Boosted Atazanavir Plus Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naïve Women
Brief Title: Safety and Efficacy of E/C/F/TDF Versus RTV-Boosted ATV Plus FTC/TDF in HIV-1 Infected, Antiretroviral Treatment-Naive Women
Acronym: WAVES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-236-0128; 2012-003708-11 (EudraCT Number)
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; HIV; Treatment-Naive; Women; WAVES
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Atazanavir Sulfate; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- E/C/F/TDF (Experimental): E/C/F/TDF + ATV placebo + RTV placebo + FTC/TDF placebo
  Interventions: Drug: E/C/F/TDF; Drug: ATV Placebo; Drug: RTV Placebo; Drug: FTC/TDF Placebo
- ATV + RTV+ FTC/TDF (Active Comparator): ATV + RTV + FTC/TDF + E/C/F/TDF placebo
  Interventions: Drug: ATV; Drug: RTV; Drug: FTC/TDF; Drug: E/C/F/TDF Placebo
- Open-Label Extension Phase (Experimental): After 48 weeks of blinded treatment, participants will continue to take blinded study drug for 12 weeks and return for an unblinding visit at Week 60. Participants who are virologically suppressed at Week 48 during the double-blinded treatment phase will have the option to enter the open-label extension phase. Participants randomized to the E/C/F/TDF arm will continue to receive open-label E/C/F/TDF and participants randomized to the ATV+ RTV + FTC/TDF arm will be re-randomized to receive either open-label elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) or open-label ATV + RTV+ FTC/TDF.
  Interventions: Drug: E/C/F/TDF; Drug: ATV; Drug: RTV; Drug: FTC/TDF; Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TDF — 150/150/200/300 mg FDC tablet administered orally with food once daily
  Other Names: Stribild®
  Arms: E/C/F/TDF; Open-Label Extension Phase
Drug: ATV — 300 mg capsule administered orally with food once daily
  Other Names: Reyataz®
  Arms: ATV + RTV+ FTC/TDF; Open-Label Extension Phase
Drug: RTV — 100 mg tablet administered orally with food once daily
  Other Names: Norvir®
  Arms: ATV + RTV+ FTC/TDF; Open-Label Extension Phase
Drug: FTC/TDF — 200/300 mg tablet administered orally with food once daily
  Other Names: Truvada®
  Arms: ATV + RTV+ FTC/TDF; Open-Label Extension Phase
Drug: E/C/F/TDF Placebo — Tablet administered orally with food once daily
  Arms: ATV + RTV+ FTC/TDF
Drug: ATV Placebo — Tablet administered orally with food once daily
  Arms: E/C/F/TDF
Drug: RTV Placebo — Capsule administered orally with food once daily
  Arms: E/C/F/TDF
Drug: FTC/TDF Placebo — Tablet administered orally with food once daily
  Arms: E/C/F/TDF
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally with food once daily
  Other Names: Genvoya®
  Arms: Open-Label Extension Phase

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a regimen containing elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF) versus ritonavir (RTV)-boosted atazanavir (ATV/r) plus emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) in HIV-1 infected, antiretroviral treatment-naive adult women.

ELIGIBILITY:
Key Inclusion Criteria:

* Female (at birth), age ≥ 18 years
* Ability to understand and sign a written informed consent form
* Plasma HIV-1 RNA levels ≥ 500 copies/mL
* No prior use of any approved or investigational antiretroviral drug for any length of time
* Screening genotype report must show sensitivity to emtricitabine (FTC), tenofovir disoproxil fumarate (TDF) and atazanavir (ATV) boosted with ritonavir (RTV)
* Normal ECG
* Adequate renal function: Estimated glomerular filtration rate ≥ 70 mL/min according to the Cockcroft Gault formula
* Hepatic transaminases ≤ 5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN
* Women of childbearing potential must agree to utilize protocol recommended contraception methods or be non-heterosexually active, or practice sexual abstinence from screening throughout the duration of the study period and for 30 days following the last dose of study drug
* Women who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing.

Key Exclusion Criteria:

* A new AIDS defining condition diagnosed within the 30 days
* Females receiving drug treatment for Hepatitis C, or females who are anticipated to receive treatment for Hepatitis C during the course of the study
* Females experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Have an implanted defibrillator or pacemaker
* Have an ECG pulse rate interval ≥ 220 msec
* Current alcohol or substance use which may potentially interfere with the female's study compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Participation in any other clinical trial without prior approval
* Any other clinical condition or prior therapy that would make the female unsuitable for the study or unable to comply with the dosing requirements
* Females receiving ongoing therapy with any disallowed medications, including drugs not to be used with elvitegravir, cobicistat, FTC, TDF, ATV, RTV; or females with any known allergies to the excipients of Stribild® tablets, Truvada® tablets, atazanavir capsules or ritonavir tablets

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2015-02-09 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (99):
- United States (41):
  - University of Southern California AIDS Clinical Trials Group, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - IDOCF/ValuhealthMD, Orlando, Florida
  - St. Joseph's Hospital Comprehensive Research Institute, Tampa, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Emory HIV/AIDS Clinical Trials Unit, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University Mercer Medicine, Macon, Georgia
  - Chatham County Health Daprtment, Savannah, Georgia
  - University of Louisville, Louisville, Kentucky
  - LSUHSC HIV Out-Patient Clinic Research, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Saint Michael's Medical Center, Newark, New Jersey
  - New Jersey Medical School, Newark, New Jersey
  - New York Hospital Queens, Flushing, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina AIDS Clinical Trials Unit, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University The Brody School of Medicine Div. of Infectious Diseases, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital- Internal General Medicine, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - UT - Physicians, Bellaire, Texas
  - AIDS Arms, Inc./Trinity Health & Wellness Center, Dallas, Texas
  - North Texas Infectious Diseases Consultants, PA, Dallas, Texas
  - Therapeutic Concepts, PA, Houston, Texas
- Belgium (3):
  - Institute of Tropical Medicine, Antwerp
  - Saint-Pierre University Hospital, Brussels
  - Hôpitaux IRIS SUD, Brussels
- Dominican Republic (2):
  - Instituto Dominicano de Estudio Virologicos - IDEV, Santo Domingo
  - Salvador B Gautier Hospital, Infectious Diseases Department, Santo Domingo
- France (4):
  - Hôpital Bichat Claude Bernard, Paris
  - Hopital Tenon, Paris
  - Maladies Infectieuses Dpt, Paris
  - Hopitaux Universitaires Strasbourg, Strasbourg
- Italy (3):
  - Department of Health Sciences - University of Milan - San Paolo Hospital, Milan
  - Luigi Sacco Hospital, Milan, Milan
  - Clinica Malattie Infettive, Azienda Ospedaliero Universitaria, Modena
- Mexico (3):
  - Hospital Civil de Guadalajara Dr Juan I Menchaca, Guadalajara, Jalisco
  - Hospital Civil de Guadalajara, Guadalajara
  - Intituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City
- Portugal (6):
  - Hospital Fernando Fonseca, Amadora
  - Hospital Dos Capuchos, Centro Hospitalar De Lisboa Central, Lisbon
  - Hospital de Santa Maria - Serviço de Doenças Infecciosas, Lisbon
  - centro Hospitalar S. João, Porto
  - Centro Hospitalar do Porto - Hospital Joaquim Urbano, Porto
  - Hospital de Santarém, Santarém
- Maternal Infants Studies Center (CEMI), San Juan, Puerto Rico
- Russia (21):
  - Republic of Altay Center for Prevention and Control of AIDS and Infectious Diseases, Barnaul
  - GUZ "Irkutsk Regional Center for Prevention and Control of AIDS and Infectious Diseases, Irkutsk
  - Khabarovsk Territorial Center for Prevention and Control of AIDS and Infectious Diseases, Khabarovsk
  - State Budget Healthcare Institution "Clinical Centre for AIDS and Infectious Diseases Fight and Prevention" of Krasnodar regio Department for Healthcare, Krasnodar
  - GUZ "Krasnoyarsk Territorial Center for Prevention and Control of AIDS and Infectious Diseases", Krasnoyarsk
  - GUZ "Lipetsk Regional Center for Prevention and Control of AIDS and Infectious Diseases", Lipetsk
  - Infectious Hospital 2, Moscow
  - State Healthcare Institution Infectious Clinical Hospital #2 of Moscow City Healthcare Department, Moscow
  - GKUZ MO "Center for Prevention and Treatment of AIDS and Infectious Diseases" (Moscow Regional AIDS Center), Moscow
  - State Budget Health Institution of Nizhniy Novgorod "Nizhniy Novgorod Regional Center of prophylaxis and treatment of AIDS and Infectious Diseases, Nizhny Novgorod
  - Budgetary Medical Facility of the Orel Region "Orel Regional Center for Prevention and Control of AIDS and Infectious Diseases", Oryol
  - Perm Regional Center for Prevention and Control of AIDS and Infectious Diseases, Perm
  - St.Petersburg Center for Prevention and Control of AIDS and Infectious Diseases, In-patient Department, Saint Petersburg
  - St.Petersburg GUZ "Center for Prevention and Control of AIDS and Infectious Diseases", Out-patient Department, Saint Petersburg
  - Saint-Petersburg GUZ "Clinical Infectious Hospital named after S.P.Botkin", Saint Petersburg
  - Federal State Budgetary Institution "Republic Clinical Infectious Hospital", Saint Petersburg
  - Saratov Regional Centre for Treatment and Prevention of AIDS and Infectious Diseases, Saratov
  - Volgograd Regional Center for Prevention and Control of AIDS and Infectious Diseases, Volgograd
  - GUZ "Voronezh Regional Center for Prevention and Control of AIDS and Infectious Diseases", Voronezh
  - Sverdlovsk Regional Center for Prevention and control of AIDS and Infectious Diseases, Yekaterinburg
  - "Infectious Diseases Center", LLC, Коltsovo
- Thailand (5):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok
  - Department of Preventive and Social Medicine, Faculty of Medicine, Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Bamrasnaradura lnfectious Disease Institute, Nonthaburi
- Joint Clinical Research Centre, Kampala, Uganda
- United Kingdom (9):
  - Barts Healthe NHS Trust, London
  - Homerton University Hospital NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Queen Elizabeth Hospital, South London Healthcare NHS Trust, London
  - Kings College London, London
  - St George's Healthcare NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Mortimer Market Centre and Central and North West London NHS Foundation Trust, London
  - Royal Berkshire NHS Foundation Trust, Reading

REFERENCES:
- [Result] Squires K, Kityo C, Hodder S, Johnson M, Voronin E, Hagins D, Avihingsanon A, Koenig E, Jiang S, White K, Cheng A, Szwarcberg J, Cao H. Integrase inhibitor versus protease inhibitor based regimen for HIV-1 infected women (WAVES): a randomised, controlled, double-blind, phase 3 study. Lancet HIV. 2016 Sep;3(9):e410-e420. doi: 10.1016/S2352-3018(16)30016-9. Epub 2016 May 27. PMID 27562742
- [Result] Hodder S, Squires K, Gathe J, Kityo C, Supparatpinyo K, Moshkovich G, et al. Elvitegravir (EVG)/cobicistat (COBI)/emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) is superior to ritonavir (RTV)-boosted atazanavir (ATV) plus FTC/TDF in treatment-naive women with HIV-1 infection (WAVES study). Presented at Interscience Conference on Antimicrobial Agents and Chemotherapy and International Congress of Chemotherapy and Infection (ICAAC/ICC) 2015; September 17-21; San Diego, CA.
- [Result] Squires K, Kityo C, Hodder S, Hagins D, Avihingsanon A, Plotnikova Y, et al. Elvitegravir (EVG)/cobicistat (COBI)/emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) is superior to ritonavir (RTV)-boosted atazanavir (ATV) plus FTC/TDF in treatment-naive women with HIV-1 infection (WAVES study). Poster no. MOLBPE08. Presented at 8th International Antiviral Society (IAS) Conference on HIV Pathogenesis, Treatment and Prevention, 2015; 19-22 July, Vancouver, BC, Canada.
- [Result] Hodder S, Kityo C, Koenig E, Mussini C, Post F, Romanova S, et al. Genotypic analysis of the global clinical trial of treatment-naive women. Abstract 16. Presented at 5th International Workshop on HIV & Women, 2015; 21-22 February, Seattle, WA.
- [Result] Squires K, Hodder S, Kityo C, Clumeck N, Johnson M, Plotnikova Y, et al. Enrollment in the Women's Antiretroviral Efficacy and Safety study (WAVES), a Phase 3 global study assessing antiretroviral regimen in treatment-naive women. Abstract 54. Presented at 5th International Workshop on HIV & Women, 2015; 21-22 February, Seattle, WA.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, Dominican Republic, Thailand, and Uganda. The first participant was screened on 24 October 2012. The last study visit occurred on 06 September 2018.
Pre-assignment Details: 810 participants were screened.
Groups:
- Double-Blind STB to Open-Label STB: Double-Blind (DB) Phase: Stribild® (STB; elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate; E/C/F/TDF) 150/150/200/300 mg fixed-dose combination (FDC) + atazanavir (ATV) placebo + ritonavir (RTV) placebo + Truvada® (TVD; emtricitabine/tenofovir disoproxil fumarate; FTC/TDF) placebo orally once daily with food for 48 weeks
  Open-Label Extension (OLE) Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to receive open-label STB FDC orally once daily with food for 48 weeks.
- Double-Blind ATV+RTV+TVD: Double-Blind Phase: ATV 300 mg + RTV 100 mg + TVD (200/300 mg) FDC + STB placebo orally once daily with food for 48 weeks
- Double-Blind ATV+RTV+TVD to Open-Label GEN: Double-Blind Phase: ATV 300 mg + RTV 100 mg + TVD (200/300 mg) FDC + STB placebo orally once daily with food for 48 weeks
  Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and receive open-label (OL) Genvoya® (GEN; elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide; E/C/F/TAF) 150/150/200/10 mg FDC orally once daily with food for 48 weeks.
- Double-Blind ATV+RTV+TVD to Open-Label ATV+RTV+TVD: Double-Blind Phase: ATV 300 mg + RTV 100 mg + TVD (200/300 mg) FDC + STB placebo orally once daily with food for 48 weeks
  Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and recieve open-label ATV 300 mg + RTV 100 mg + TVD 200/300 mg FDC orally once daily with food for 48 weeks.
Period: Double-Blind Phase
Arm/Group | Double-Blind STB to Open-Label STB | Double-Blind ATV+RTV+TVD | Double-Blind ATV+RTV+TVD to Open-Label GEN | Double-Blind ATV+RTV+TVD to Open-Label ATV+RTV+TVD
Started | 293 | 290 | 0 | 0
Completed | 260 | 249 | 0 | 0
Not Completed | 33 | 41 | 0 | 0
Not completed — Lost to Follow-up | 12 | 16 | 0 | 0
Not completed — Adverse Event | 3 | 10 | 0 | 0
Not completed — Withdrew Consent | 8 | 5 | 0 | 0
Not completed — Non-Compliance with Study Drug | 4 | 5 | 0 | 0
Not completed — Pregnancy | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Randomized but Not Treated | 4 | 4 | 0 | 0
Period: Open-Label Extension Phase
Arm/Group | Double-Blind STB to Open-Label STB | Double-Blind ATV+RTV+TVD | Double-Blind ATV+RTV+TVD to Open-Label GEN | Double-Blind ATV+RTV+TVD to Open-Label ATV+RTV+TVD
Started (14 participants did not enter the OLE STB arm.) | 246 | 0 (Participants either entered the OL GEN arm or OL ATV+RTV+TVD arm.) | 159 (159 participants entered from the DB ATV+RTV+TVD arm.) | 53 (53 participants entered from the DB ATV+ RTV + TVD arm.)
Completed | 231 | 0 | 148 | 48
Not Completed | 15 | 0 | 11 | 5
Not completed — Lost to Follow-up | 6 | 0 | 2 | 2
Not completed — Withdrew Consent | 4 | 0 | 4 | 1
Not completed — Adverse Event | 3 | 0 | 0 | 1
Not completed — Death | 2 | 0 | 1 | 0
Not completed — Non-Compliance with Study Drug | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were randomized and received at least one dose of study drug.
Groups:
- Double-Blind STB to Open-Label STB: Double-Blind Phase: STB 150/150/200/300 mg FDC + ATV placebo + RTV placebo + TVD placebo orally once daily with food for 48 weeks
  Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to receive open-label STB FDC orally once daily with food for 48 weeks.
- Double-Blind ATV+RTV+TVD to OL GEN or OL ATV+ RTV+TVD: Double-Blind Phase: ATV 300 mg + RTV 100 mg + TVD (200/300 mg) FDC + STB placebo orally once daily with food for 48 weeks
  Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and either receive open-label GEN 150/150/200/10 mg FDC or open-label ATV 300 mg + RTV 100 mg + TVD 200/300 mg FDC orally once daily with food for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Double-Blind STB to Open-Label STB | Double-Blind ATV+RTV+TVD to OL GEN or OL ATV+ RTV+TVD | Total
Number analyzed (Participants) | 289 | 286 | 575
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10.1) | 36 (9.7) | 36 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289 | 286 | 575
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 17 | 26
  Black | 143 | 133 | 276
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  White | 128 | 119 | 247
  Other | 9 | 15 | 24
  Not Permitted | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 24 | 44
  Not Hispanic or Latino | 269 | 262 | 531
  Not Permitted | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 101 | 91 | 192
  United States | 59 | 60 | 119
  United Kingdom | 8 | 12 | 20
  Thailand | 9 | 15 | 24
  Portugal | 8 | 13 | 21
  Belgium | 3 | 5 | 8
  Dominican Republic | 6 | 13 | 19
  Italy | 4 | 1 | 5
  Mexico | 3 | 1 | 4
  Uganda | 87 | 74 | 161
  France | 1 | 1 | 2
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 376 (199.6) | 385 (210.2) | 381 (204.8)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 220 | 214 | 434
  > 100,000 to ≤400,000 copies/mL | 44 | 50 | 94
  > 400,000 copies/mL | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 of the Double-Blind Phase as Determined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 of the double-blind phase was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Intent-to-Treat (ITT) Analysis Set (randomized and received at least one dose of study drug) were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Double-Blind STB: Double-Blind Phase: STB 150/150/200/300 mg FDC + ATV placebo + RTV placebo + TVD placebo orally once daily with food for 48 weeks
- Double-Blind ATV+RTV+TVD: Double-Blind Phase: ATV 300 mg boosted with RTV 100 mg + TVD (200/300 mg) FDC + E/C/F/TDF placebo once daily for 48 weeks
Arm/Group | Double-Blind STB | Double-Blind ATV+RTV+TVD
Number analyzed (Participants) | 289 | 286
percentage of participants | 87.2 | 80.8
Statistical Analysis 1: Comparison: Double-Blind STB vs Double-Blind ATV+RTV+TVD; Test type: Non-Inferiority or Equivalence — The null hypothesis was that the STB group was at least 12% worse than the ATV+RTV+TVD group with respect to the percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 (response rate as defined by the snapshot analysis algorithm). The alternative hypothesis was that the STB group was less than 12% worse than the ATV+RTV+TVD group; Difference in proportions = 6.5, 95.2% CI 2-sided [0.4 to 12.6] — Difference in percentages of virologic success and its 95.2% confidence interval (CI) were calculated based on baseline HIV-1 RNA and race stratum-adjusted Mantel-Haenszel (MH) proportion
Statistical Analysis 2: Comparison: Double-Blind STB vs Double-Blind ATV+RTV+TVD; If noninferiority of STB versus ATV+RTV+TVD was established, the same 95.2% CI used in evaluating noninferiority was used to evaluate superiority. The baseline HIV-1 RNA and race stratum-stratified, 2-sided CMH test was also used to assess superiority as a secondary assessment; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel; P-value comparing virologic success was from the CMH test stratified by baseline HIV-1 RNA and race strata; Difference in proportions = 6.5, 95.2% CI 2-sided [0.4 to 12.6] — Difference in percentages of virologic success and its 95.2% CI were calculated based on baseline HIV-1 RNA and race stratum-adjusted MH proportion. If the lower bound of the CI was > 0, superiority of STB over ATV+RTV+TVD was established

2. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48 of the Double-Blind Phase
Time Frame: Baseline; Week 48
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Double-Blind STB | Double-Blind ATV+RTV+TVD
Number analyzed (Participants) | 263 | 243
cells/μL | 221 (165.1) | 212 (176.8)

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 for the STB Group as Determined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the ITT Analysis Set who received STB through 96 weeks were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- ALL STB: Double-Blind Phase: STB 150/150/200/300 mg FDC + ATV placebo + RTV placebo + TVD placebo orally once daily with food for 48 weeks
  Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had option to receive open-label STB FDC orally once daily with food for 48 weeks.
Arm/Group | ALL STB
Number analyzed (Participants) | 278
Percentage of participants | 84.5 [79.7 to 88.6]

4. Secondary Outcome: Percentage of Participants Receiving STB or ATV+RTV+TVD With HIV-1 RNA < 50 Copies/mL at Week 48 of the Open-Label Extension Phase
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 of the open-label phase was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Open-Label Extension Week 48
Population: Participants in the OLE ITT Analysis Set were analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- Open-Label GEN: Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and receive open-label GEN 150/150/200/10 mg FDC orally once daily with food for 48 weeks.
- Open-Label ATV+RTV+TVD: Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and receive open-label ATV 300 mg + RTV 100 mg + TVD 200/300 mg FDC orally once daily with food for 48 weeks.
Arm/Group | Open-Label GEN | Open-Label ATV+RTV+TVD
Number analyzed (Participants) | 159 | 53
Percentage of participants | 94.3 | 86.8

5. Secondary Outcome: Change in CD4+ Cell Count at Week 48 of the Open-Label Extension Phase
Time Frame: Baseline; Open-Label Extension Week 48
Population: Participants in the OLE ITT Analysis Set with available on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/uL
Groups:
- Open-Label STB: Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to receive open-label STB FDC orally once daily with food for 48 weeks.
- Open-Label ATV + RTV + TVD: Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and receive open-label ATV 300 mg + RTV 100 mg + TVD 200/300 mg FDC orally once daily with food for 48 weeks.
Arm/Group | Open-Label STB | Open-Label GEN | Open-Label ATV + RTV + TVD
Number analyzed (Participants) | 239 | 151 | 49
cells/uL | 265 (190.4) | 35 (137.5) | 49 (204.8)

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date plus 30 days including DB phase and OLE phase (maximum duration: ALL STB (DB STB and OL STB) = 239.9 weeks; DB ATV+RTV+TVD = 90.6 weeks; DB ATV+ RTV+TVD to OL GEN = 191.3 weeks; DB ATV+RTV+TVD to OL ATV+RTV+TVD = 102.0 weeks)
Description: Adverse events reported included randomized participants who received at least 1 dose of any drug in either DB phase or OLE phase.
Groups:
- Double-Blind: STB: Double-Blind Phase: STB 150/150/200/300 mg FDC + ATV placebo + RTV placebo + TVD placebo orally once daily with food for 48 weeks
- Double-Blind: ATV+RTV+TVD: Double-Blind Phase: ATV 300 mg + RTV 100 mg + TVD (200/300 mg) FDC + STB placebo orally once daily with food for 48 weeks
- DB STB to OL STB: Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to receive open-label STB FDC orally once daily with food for 48 weeks.
- DB ATV+RTV+TVD to OL GEN: Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and receive open-label GEN 150/150/200/10 mg FDC orally once daily with food for 48 weeks.
- DB ATV+RTV+TVD to OL ATV+RTV+TVD: Open-Label Extension Phase: After 48 weeks of blinded treatment participants continued on the blinded treatment for 12 weeks and returned for an unblinding visit at Week 60. Participants who were virologically suppressed at Week 48 during the double-blind phase had the option to be re-randomized and recieve open-label ATV 300 mg + RTV 100 mg + TVD (200/300 mg) FDC orally once daily with food for 48 weeks.
Arm/Group | Double-Blind: STB | Double-Blind: ATV+RTV+TVD | DB STB to OL STB | DB ATV+RTV+TVD to OL GEN | DB ATV+RTV+TVD to OL ATV+RTV+TVD
Serious Adverse Events (participants affected / at risk) | 25/289 | 29/286 | 13/246 | 12/159 | 4/53
Other Adverse Events (participants affected / at risk) | 176/289 | 194/286 | 118/246 | 68/159 | 20/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: STB (N=289) | Double-Blind: ATV+RTV+TVD (N=286) | DB STB to OL STB (N=246) | DB ATV+RTV+TVD to OL GEN (N=159) | DB ATV+RTV+TVD to OL ATV+RTV+TVD (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bone tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 1 | 3 | 2
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: STB (N=289) | Double-Blind: ATV+RTV+TVD (N=286) | DB STB to OL STB (N=246) | DB ATV+RTV+TVD to OL GEN (N=159) | DB ATV+RTV+TVD to OL ATV+RTV+TVD (N=53)
Anaemia (Blood and lymphatic system disorders) | 11 | 14 | 18 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 17 | 9 | 1 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 15 | 19 | 6 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 13 | 15 | 4 | 3 | 0
Nausea (Gastrointestinal disorders) | 43 | 41 | 6 | 7 | 2
Vomiting (Gastrointestinal disorders) | 28 | 17 | 3 | 4 | 0
Fatigue (General disorders) | 8 | 15 | 2 | 3 | 2
Jaundice (Hepatobiliary disorders) | 1 | 30 | 0 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 1 | 34 | 0 | 0 | 0
Influenza (Infections and infestations) | 20 | 20 | 14 | 12 | 1
Malaria (Infections and infestations) | 34 | 25 | 14 | 8 | 1
Nasopharyngitis (Infections and infestations) | 15 | 14 | 8 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 50 | 45 | 36 | 23 | 10
Urinary tract infection (Infections and infestations) | 22 | 23 | 15 | 9 | 0
Vulvovaginal candidiasis (Infections and infestations) | 21 | 20 | 15 | 6 | 4
Decreased appetite (Metabolism and nutrition disorders) | 15 | 14 | 3 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 21 | 9 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 17 | 13 | 14 | 1
Dizziness (Nervous system disorders) | 17 | 10 | 7 | 0 | 1
Headache (Nervous system disorders) | 49 | 44 | 27 | 20 | 5
Neuropathy peripheral (Nervous system disorders) | 21 | 20 | 12 | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 18 | 12 | 9 | 2

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years